CLINICAL TRIAL: NCT07330947
Title: Incidence and Risk Factors of Postoperative Chronic Pain in Patients Who Have Undergone Hallux Valgus Surgery in the UC-Christus Clinical Hospital
Brief Title: Incidence and Risk Factors of Postoperative Chronic Pain in Patients Who Have Undergone Hallux Valgus Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, María Francisca Elgueta Le-beuffe, MD Anesthesiologist and Associate Professor, Pontificia Universidad Catolica de Chile
Other Study IDs: 240930004
Record Dates: First submitted 2025-11-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Chronic Pain; Hallux Valgus Surgery
Keywords: Hallux Valgus surgery; postoperative chronic pain; risk factors; brief pain inventory
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the incidence and risk factors of postoperative chronic pain in adult patients who have undergone Hallux Valgus surgery (between january 2021 and december 2024). This will be assesed through scales and medical records information.

The main questions to be answered are:

* How many patients who have undergone Hallux Valgus surgery are experiencing postoperative chronic pain.
* What factors are there present in those who do experience chronic pain after surgery.

After accepting the informed consent, participants will be asked to answer a Brief Pain Inventory Scale and a Risk Factor Questionnaire for Postoperative Chronic Pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent Hallux Valgus surgery at various centers within the UC Christus network from January 2021 to April 2024.

Exclusion Criteria:

* Patients who had difficulty responding to follow-up from the UC Christus health network Pain Unit and/or who do not answer the telephone call

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a descriptive cross-sectional study involving 350 patients who underwent Hallux Valgus surgery at a Clinical Hospital from January 2021 to April 2024.
  The study includes patients who underwent Hallux Valgus surgery within the UC Christus Health Network.
  The telephone records of patients who meet the inclusion criteria will be obtained from the Orthopedics Service database, in adherence to the UC Christus clinical data protection policy.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of Chronic Postoperative Pain (CPOP) following Hallux Valgus surgeries | "Day 1" The outcome measure will be recorded on day 1, when the patient has agreed to the informed consent and to answer the questionnaire.
  The main outcome (chronic pain related to Hallux Valgus surgeries) will be assessed through the Brief Pain Inventory scale:
  * Pain intensity: Moderate (Visual Analog Scale 5 - 7) or severe pain (Visual Analog Scale 8 - 10).
  * Time: over 3 months.
  * Pain description: pain is anatomically located where the Hallux Valgus surgery has taken place.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile